CLINICAL TRIAL: NCT04251234
Title: Light at Night Study
Acronym: LAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID shutdown
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Helen Burgess, Professor of Psychiatry, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00173528
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Disorder; Light Sensitivity
Keywords: Circadian; Light Intensity
MeSH Terms: conditions — Bipolar Disorder; Photophobia

STUDY DESIGN:
Masking Description: There is no masking. The dim light (<1 lux) condition is first, followed by the room light (~30 lux) condition. Participants are aware of this condition order.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (Experimental): * No co-morbid medical or psychiatry diagnoses
  * No family history of mental illness
  * No current medication use
  * Non-smoking
  Interventions: Other: Light intensity, ~30 lux; Other: Baseline light intensity, <1 lux
- Bipolar I disorder (Experimental): * Clinical diagnosis of Bipolar I disorder
  * Can be (not required, not exclusionary) taking lithium and/or sodium valproate and/or antidepressants
  * Can be (not required, not exclusionary) light smokers
  Interventions: Other: Light intensity, ~30 lux; Other: Baseline light intensity, <1 lux

INTERVENTIONS:
Other: Light intensity, ~30 lux — ~30 lux compared to very dim light baseline condition <1 lux
Other: Baseline light intensity, <1 lux — Very dim light condition

SUMMARY:
The purpose of this mechanistic study is to examine light sensitivity (melatonin suppression) in people with bipolar depression I, and compare it to healthy controls. This is not a treatment study.

DETAILED DESCRIPTION:
The bipolar disorder I and healthy control arms are recruited from the existing Heinz C. Prechter Bipolar Research Program at the University of Michigan.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30 kg/m2
* Appropriate sleep schedules according to study staff. Sleep schedule is self-reported and confirmed through a sleep diary
* Healthy eyes as ascertained by eye exam at University of Michigan Kellogg Eye Center
* Willing and able to maintain stable sleep schedule during study.
* Participants will be breathalyzed and undergo urine drugs screens at every lab visit
* Acknowledge and understand that participants cannot drive themselves home after certain lab visits. Note that the research team will provide a travel stipend of $10 per visit to offset potential rideshare/taxi costs

Exclusion Criteria:

* Color blindness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Melatonin levels | Up to approximately 6 weeks
  Melatonin will be reported as an average percentage of suppression in the ~30 lux condition as compared to <1 lux

CONTACTS AND LOCATIONS:
Overall Officials: Helen Burgess, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No